CLINICAL TRIAL: NCT00196144
Title: Far Field Sensing Test Study in Patients With Implanted Cardiac Dual Chamber Pacemakers
Brief Title: FFS - Far Field Sensing Test Study in Cardiac Dual Chamber Pacemakers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GE IDE No. P00202
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Optimization of the postventricular atrial blanking period to avoid far-field R-wave sensing.
  Interventions: Device: Individualized Programming of PVAB
- 2 (Experimental): Programming of the nominal setting for the post-ventricular atrial blanking period (100 ms)
  Interventions: Device: Nominal PVAB

INTERVENTIONS:
Device: Individualized Programming of PVAB — Performance of a test to detect far-field R-wave sensing
  Arms: 1
Device: Nominal PVAB — nominal pacemaker settings
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of individual adjustment of the postventricular atrial blanking period in avoiding inappropriate mode switch of dual chamber pacemakers.

DETAILED DESCRIPTION:
Far-field R-wave sensing (FFS) in the atrial channel of dual chamber pacemakers is a relevant source for inappropriate mode switch from the DDD mode to the DDI or VDI mode. Inappropriate loss of atrioventricular synchrony due to false positive mode switch is hemodynamically disadvantageous, may induce atrial tachyarrhythmias, can lead to pacemaker syndrome, and impairs the reliability of pacemaker Holter data. The aim of the study is to determine whether individual adjustment of the postventricular atrial blanking period (PVAB) based on an additional test is effective in avoiding inappropriate mode switch due to FFS when compared to standard programming of the PVAB

ELIGIBILITY:
Inclusion Criteria:

* Indication for dual chamber pacing
* Implantation of an Identity DR pacemaker (St. Jude Medical)
* Bipolar atrial pacing electrode

Exclusion Criteria:

* Heart failure NYHA III and IV
* Unstable angina pectoris
* Indication for the implantation of an ICD
* Cardiac surgery within previous 6 months
* Cardiac surgery planed for the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2002-07; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Incidence of inappropriate mode switch due to far field R-wave sensing | 3 months

SECONDARY OUTCOMES:
Incidence of inappropriate mode switch due to far field R-wave sensing in relation to the lead position | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Schmitt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Christof Kolb, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Result] Kolb C, Wille B, Maurer D, Schuchert A, Weber R, Schibgilla V, Klein N, Hummer A, Schmitt C, Zrenner B; FFS-Test Study Group. Management of far-field R wave sensing for the avoidance of inappropriate mode switch in dual chamber pacemakers: results of the FFS-test study. J Cardiovasc Electrophysiol. 2006 Sep;17(9):992-7. doi: 10.1111/j.1540-8167.2006.00545.x. PMID 16948743